CLINICAL TRIAL: NCT04205955
Title: A Randomized Trial of the Altering Intake, Managing Symptoms Intervention for Bowel Dysfunction in Rectal Cancer Survivors Compared to a Healthy Living Education Control: A Feasibility and Preliminary Efficacy Study (AIMS-RC)
Brief Title: Testing Diet Intervention Versus Non-Diet Intervention for Management of Bowel Symptoms in Rectal Cancer Survivors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: S1820; NCI-2019-04990 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1820 (Other: SWOG); SWOG-S1820 (Other: DCP); S1820 (Other: CTEP); R21CA236057 (NIH); UG1CA189974 (NIH)
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Results first posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Rectal Carcinoma; Rectosigmoid Carcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (diet modification coaching, motivational messages) (Experimental): Patients receive diet modification coaching via telephone for 10 sessions over 30-60 minutes over 17 weeks. Patients also receive 3 motivational messages per week via email and/or text message beginning after session 6.
  Interventions: Dietary Supplement: Dietary Intervention; Other: Message; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (standard of care, motivational messages) (Active Comparator): Patients receive general healthy living education via telephone for 10 sessions over 30-60 minutes over 17 weeks. Patients also receive 3 motivational messages per week via email and/or text message beginning after session 6.
  Interventions: Other: Best Practice; Other: Message; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive healthy living education via phone call
  Other Names: standard of care; standard therapy
  Arms: Arm II (standard of care, motivational messages)
Dietary Supplement: Dietary Intervention — Receive diet modification coaching via phone call
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Arm I (diet modification coaching, motivational messages)
Other: Message — Receive motivational messages via email and/or text message
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how a diet intervention works in improving bowel dysfunction symptoms related in colon or rectal cancer survivors. Changing a diet may be helpful in reducing the severity of bowel symptoms, including diarrhea and constipation, and improve quality of life in colon or rectal cancer survivors and help doctors learn how to help patients better in the future.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare total bowel function score, as measured by the Memorial Sloan-Kettering Cancer Center Bowel Function Instrument (BFI), at 18 weeks post-randomization between the intervention and attention control arms.

EXPLORATORY OBJECTIVES:

I. To compare total bowel function score at 26 weeks post-randomization between the intervention and attention control arms.

II. To compare bowel function subscale scores (dietary, urgency, frequency), as measured by the BFI at both 18- and 26- weeks post-randomization between the intervention and attention control arms.

III. To compare lower anterior resection syndrome (LARS) scores (for anastomosis participants only), quality of life, and dietary quality at both 18- and 26- weeks post-randomization between the intervention and attention control arms.

IV. To compare motivation, self-efficacy, and positive/negative affect at both 18- and 26- weeks post-randomization between the intervention and attention control arms.

V. To assess study feasibility, adherence, retention, and acceptability at both 18 and 26 weeks post-randomization.

VI. To explore variation in primary and exploratory study outcomes according to sex, and to investigate whether intervention effects on the primary outcome differ across subgroups defined by sex.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive diet modification coaching via telephone for 10 sessions over 30-60 minutes over 17 weeks. Patients also receive 3 motivational messages per week via email and/or text message beginning after session 6.

ARM II: Patients receive general healthy living education via telephone for 10 sessions over 30-60 minutes over 17 weeks. Patients also receive 3 motivational messages per week via email and/or text message beginning after session 6.

After completion of study, patients are followed up at 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* PRIOR TO STEP 1 REGISTRATION:
* Patients must have prior history of rectosigmoid colon cancer or rectal cancer
* Patients must have a post-surgical permanent ostomy or anastomosis
* Patient's last date of treatment for rectal cancer (any surgery, chemotherapy, radiation therapy) must be at least 6 months prior to registration and not more than 24 months prior to registration
* Anastomosis patients must have low anterior resection syndrome (LARS) score of 21-42 (minor to major symptoms) within 5 calendar days prior to registration
* Patient must have completed all baseline questionnaires within 5 days prior to registration
* Patients must be able to read, write and speak English. Study materials and telephone calls are only available in English
* Patients with a prior malignancy or concurrent malignancy that is currently not being treated, whose natural history or treatment (in the opinion of the treating physician) does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients who are currently undergoing treatment for another cancer will have a different symptom profile than what this study is targeting and are not eligible
* Patients who have been diagnosed with inflammatory bowel disease (IBD), such as ulcerative colitis or Crohn's disease, are not eligible
* PRIOR TO STEP 2 REGISTRATION:
* Patient must meet all eligibility criteria for step 1
* Patient must have successfully completed ("pass") the run-in period, as per email notification from the University of Arizona
* Patient must be registered to step 2 no more than 40 days after step 1 registration. If day 40 falls on a weekend or holiday, the limit may be extended to the next working day
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, Principal Investigator — SWOG Cancer Research Network
Locations (226):
- United States (225):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - John Fitzgerald Kennedy Medical Center, Atlantis, Florida
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Savio, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Joseph Regional Medical Center, Lewiston, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - HaysMed University of Kansas Health System, Hays, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Indian Creek Campus, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Maine Medical Partners Surgical Care, Portland, Maine
  - MMP Surgical Care Casco Bay, Portland, Maine
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Beaumont Hospital - Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Beaumont Hospital - Farmington Hills, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - McLaren-Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Mid-Michigan Medical Center - Midland, Midland, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - M D Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Valley Health / Winchester Medical Center, Winchester, Virginia
  - Skagit Valley Hospital Regional Cancer Care Center, Mount Vernon, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Olympic Medical Cancer Care Center, Sequim, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- FHP Health Center-Guam, Tamuning, Guam

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 95 participants were randomly assigned; 48 on the attention control arm and 47 on the intervention arm. Reasons for ineligibility include not completing run-in, withdraw of consent, and disease progression.
Period: Overall Study
Arm/Group | Arm I (Diet Modification Coaching, Motivational Messages) | Arm II (Standard of Care, Motivational Messages)
Started | 47 | 48
Completed | 47 | 48
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Diet Modification Coaching, Motivational Messages) | Arm II (Standard of Care, Motivational Messages) | Total
Number analyzed (Participants) | 47 | 46 | 93
Age, Continuous [Median (Full Range); unit: years] | 54.6 [30.3 to 81.2] | 56.9 [26.7 to 86.7] | 55.2 [26.7 to 86.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 51
  Male | 20 | 22 | 42
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 2 | 2 | 4
  Asian | 4 | 3 | 7
  Black or African American | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Unknown | 2 | 0 | 2
  White | 38 | 39 | 77
Ethnicity [Count of Participants; unit: Participants]
  Hispanic | 3 | 4 | 7
  Non-Hispanic | 42 | 40 | 82
  Unknown | 2 | 2 | 4
Highest Level of Education [Count of Participants; unit: Participants]
  Did not complete high school | 2 | 0 | 2
  Completed high school/GED/vocational/secretarial/business | 7 | 10 | 17
  Any college | 23 | 24 | 47
  Any graduate school | 15 | 12 | 27
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 27.3 [17.1 to 52.3] | 27.6 [19.1 to 66.3] | 27.3 [17.1 to 66.3]
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  <18.5 kg/m^2 (Underweight) | 2 | 0 | 2
  18.5-<25 kg/m^2 (Normal weight) | 13 | 12 | 25
  25-<30 kg/m^2 (Overweight) | 16 | 18 | 34
  >=30 kg/m^2 (Obese) | 16 | 16 | 32
Smoking Status [Count of Participants; unit: Participants]
  Current | 1 | 1 | 2
  Former | 9 | 15 | 24
  Never | 35 | 28 | 63
  Unknown | 2 | 2 | 4
Current Marital Status [Count of Participants; unit: Participants]
  Divorced | 7 | 6 | 13
  Married or partnered | 34 | 31 | 65
  Single | 5 | 7 | 12
  Widowed | 1 | 2 | 3
Any Change in Marital Status Since Diagnosis [Count of Participants; unit: Participants]
  Yes | 1 | 5 | 6
  No | 46 | 41 | 87
Adjusted Diet because of Surgery/ostomy [Count of Participants; unit: Participants]
  Yes | 35 | 35 | 70
  No | 12 | 11 | 23
Time to Comfort with Diet after your Surgery/ostomy [Count of Participants; unit: Participants]
  Less than 1 month | 6 | 6 | 12
  1 to 12 months | 15 | 12 | 27
  More than 12 months | 3 | 3 | 6
  I am still not comfortable | 22 | 25 | 47
  Not Answered | 1 | 0 | 1
Time Since Diagnosis [Median (Full Range); unit: months] | 23.6 [8.1 to 56.7] | 22.3 [10.5 to 36.0] | 23.3 [8.1 to 56.7]
Type of Cancer [Count of Participants; unit: Participants]
  Rectal | 39 | 38 | 77
  Rectosigmoid colon | 8 | 7 | 15
  Other | 0 | 1 | 1
Prior Treatment: Chemotherapy [Count of Participants; unit: Participants]
  Yes | 41 | 42 | 83
  No | 6 | 4 | 10
Prior Treatment: Radiation Therapy [Count of Participants; unit: Participants]
  Yes | 33 | 38 | 71
  No | 14 | 8 | 22
Prior Surgery: Anastomosis [Count of Participants; unit: Participants]
  Yes | 24 | 16 | 40
  No | 23 | 30 | 53
Prior Surgery: Ostomy [Count of Participants; unit: Participants]
  Yes | 6 | 9 | 15
  No | 41 | 37 | 78
Prior Surgery: Temporary Ostomy and Re-anastomosis [Count of Participants; unit: Participants]
  Yes | 17 | 21 | 38
  No | 30 | 25 | 55
Time Since Surgery [Median (Full Range); unit: months] | 15.9 [6.2 to 51.9] | 13.6 [6.4 to 29.7] | 14.0 [6.2 to 51.9]
Type of Low Anterior Resection Surgery [Count of Participants; unit: Participants]
  Abdominoperineal resection | 5 | 10 | 15
  Low anterior resection | 42 | 34 | 76
  Sigmoid colectomy | 0 | 2 | 2
LAR Syndrome (LARS) Burden [Count of Participants; unit: Participants] — LAR = Lower Anterior Resection. Valid for anastomosis patients only. Score range 0-42: No LARS (0-20), Minor LARS (21-29), Major LARS (30-42).
  Participants
    Minor LARS | 6 | 6 | 12
    Major LARS | 35 | 31 | 66
    Not applicable, ostomy | 6 | 9 | 15
Zubrod Performance Status [Count of Participants; unit: Participants] — A performance status of 0 is defined as fully active, able to carry on all pre-disease performance without restriction.
  A performance status of 1 is defined as restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  A performance status of 2 is defined as ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    0 | 37 | 31 | 68
    1 | 8 | 14 | 22
    2 | 1 | 0 | 1
    Missing | 1 | 1 | 2
Current Medication: Antibiotics [Count of Participants; unit: Participants]
  Yes | 0 | 2 | 2
  No | 47 | 44 | 91
Current Medication: Antidiarrheal Medications [Count of Participants; unit: Participants]
  Yes | 15 | 13 | 28
  No | 32 | 33 | 65
Current Medication: Medication for Constipation [Count of Participants; unit: Participants]
  Yes | 11 | 10 | 21
  No | 36 | 36 | 72
Current Medication: Probiotics [Count of Participants; unit: Participants]
  Yes | 11 | 7 | 18
  No | 36 | 39 | 75
Used Alternative Therapies for Bowel Issues in Past 5 Months [Count of Participants; unit: Participants] — Includes meditation, mindfulness therapy, acupuncture, or other alternative therapies
  Participants
    Yes | 5 | 4 | 9
    No | 42 | 42 | 84
AJCC clinical stage at diagnosis: T Stage [Count of Participants; unit: Participants] — Tx: Unmeasured tumor T1: Tumor is only in the inner layer of the bowel T2: Tumor has grown into the muscle layer of the bowel wall T3: Tumor has grown into the outer lining of the bowel wall T4: Tumor has grown through the bowel wall into near by organs
  Participants
    T1 | 4 | 3 | 7
    T2 | 9 | 6 | 15
    T3 | 33 | 31 | 64
    T4 | 1 | 5 | 6
    TX | 0 | 1 | 1
AJCC Clinical Stage at Diagnosis: N Stage [Count of Participants; unit: Participants] — NX: Cancer in nearby lymph nodes cannot be measured. N0: There is no cancer in nearby lymph nodes. N1: One near by lymph node contains cancer. N2: Two near by lymph nodes contain cancer.
  Participants
    N0 | 18 | 13 | 31
    N1 | 14 | 21 | 35
    N2 | 12 | 10 | 22
    NX | 3 | 2 | 5
AJCC Clinical Stage at Diagnosis: M Stage [Count of Participants; unit: Participants] — MX: Metastasis cannot be measured. M0: Cancer has not spread to other parts of the body. M1: Cancer has spread to other parts of the body.
  Participants
    M0 | 41 | 42 | 83
    M1 | 2 | 0 | 2
    MX | 2 | 3 | 5
    Missing | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Bowel Function
Description: Will be measured by the Memorial Sloan-Kettering Cancer Center Bowel Function Instrument (BFI) total score. Score range 18-90. Higher scores indicate better bowel function. Will be conducted according to a modified intention-to-treat principle. Study arm differences in BFI at 18 weeks will be assessed by a linear regression model as a function of randomization assignment, BFI baseline value, and stratification factors.
Time Frame: At 18 weeks after randomization
Population: 95 total participants were randomly assigned; 47 on the intervention arm and 46 on the attention control arm. 3 patients were deemed ineligible for missing assessments and for other ineligibility criteria. This leaves 46 participants on the intervention arm and 44 on the attention control arm.
Measure: Mean (95% Confidence Interval); unit: MSK-BFI score on a scale (range 18-90)
Arm/Group | Arm I (Diet Modification Coaching, Motivational Messages) | Arm II (Standard of Care, Motivational Messages)
Number analyzed (Participants) | 46 | 44
MSK-BFI score on a scale (range 18-90) | 30.8 [29.2 to 32.4] | 29.5 [27.3 to 31.7]

2. Other Pre Specified Outcome: Bowel Function
Description: Will describe using dietary, urgency, and frequency scales. Will be assessed by a repeated measures linear regression model as a function of randomization assignment, baseline value of the outcome, stratification factors, and visit. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
Time Frame: Up to week 26
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Low Anterior Resection Syndrome (LARS)
Description: LARS will be measured using the LARS Score. Will be assessed by a repeated measures linear regression model as a function of randomization assignment, baseline value of the outcome, stratification factors, and visit. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
Time Frame: Up to week 26
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Quality of Life-Assessment
Description: Will be measured by the City of Hope-Quality of Life-Colorectal Cancer. Will be assessed by a repeated measures linear regression model as a function of randomization assignment, baseline value of the outcome, stratification factors, and visit. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
Time Frame: Up to week 26
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Dietary Quality
Description: Will be based on the Healthy Eating Index 2015. Will be assessed by a repeated measures linear regression model as a function of randomization assignment, baseline value of the outcome, stratification factors, and visit. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
Time Frame: Up to week 26
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Motivation
Description: Will be measured using a 10-item scale assessing motivation to change dietary behaviors in rectal cancer survivors. Will be assessed by a repeated measures linear regression model as a function of randomization assignment, baseline value of the outcome, stratification factors, and visit. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
Time Frame: Up to week 26
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Self-efficacy
Description: Will be measured using the Patient-Reported Outcomes Measurement Information System Self-Efficacy for Managing Symptoms - Short Form 4a. Will be assessed by a repeated measures linear regression model as a function of randomization assignment, baseline value of the outcome, stratification factors, and visit. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
Time Frame: Up to week 26
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Positive and Negative Effects
Description: Will be measured using the International Positive and Negative Affect Schedule Short Form. Will be assessed by a repeated measures linear regression model as a function of randomization assignment, baseline value of the outcome, stratification factors, and visit. Robust standard errors will be estimated via generalized estimating equations to adjust for correlation between repeated outcome measures. The dependent variables will be transformed to approximate normality as appropriate.
Time Frame: Up to week 26
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Feasibility of the Intervention
Description: Will be measured by the percentage of patients who successfully complete ("pass") the run-in period, and randomized. Accrual rates and feasibility will be summarized.
Time Frame: Up to week 26
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Adherence to the Intervention
Description: Will measure successful completion of intervention or attention control coaching calls. Adherence is defined as completing all five of sessions 1-5 and at least three of sessions 6-10 within 18 weeks after randomization. Study arm differences in adherence will be assessed by chi square tests.
Time Frame: Up to week 18
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Retention to the Intervention
Description: Will be defined by completion of follow-up assessments in step 2, including those administered at follow-up site visits and the dietary recalls. Study arm differences in retention will be assessed by chi square tests.
Time Frame: Up to week 26
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Acceptability to the Intervention
Description: Will be measured using the Acceptability of Intervention measure. Study program acceptability will be compared across arms via t-test.
Time Frame: Up to week 26
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events were not collected
Description: Adverse Events were not collected
Arm/Group | Arm I (Diet Modification Coaching, Motivational Messages) | Arm II (Standard of Care, Motivational Messages)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT04205955/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT04205955/ICF_001.pdf